CLINICAL TRIAL: NCT01366768
Title: Release of Gut Hormones After Oral Versus Intravenous Amino Acids
Brief Title: Gut Hormones After Oral Versus Intravenous Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 003
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Normal Non-fluency
Keywords: Gut hormones; Insulin secretion; Normal physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral amino acid mixture (Experimental): Oral administration of amino acid mixture in healthy volunteers
  Interventions: Other: Oral amino acid mixture
- Intravenous amino acid administration (Experimental): Intravenous infusion of amino acid mixture in healthy volunteers
  Interventions: Other: Intravenous amino acid administration

INTERVENTIONS:
Other: Oral amino acid mixture — Amino acid mixture 2,93 ml/kg
  Other Names: Amino acid mixture
  Arms: Oral amino acid mixture
Other: Intravenous amino acid administration — Amino acid mixture 2,93 ml/kg
  Other Names: Amino acid mixture
  Arms: Intravenous amino acid administration

SUMMARY:
The study hypothesis is that gut hormones are released after oral but not intravenous amino acids which result in stimulation of insulin secretion.

DETAILED DESCRIPTION:
Amino acid mixture is given orally or intravenously to match total concentrations of amino acids in healthy subjects. Samples are taken regularly for 300 min after administrations. Plasma levels of the gut hormones glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 (GLP-1)and determined and related to plasma levels of insulin and glucagon.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Diabetes
* Liver disease
* Kidney disease
* Thyroid disease

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Gut hormone secretion | 300 min

SECONDARY OUTCOMES:
Insulin secretion | 300 min

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Clinical Sciences Lund, Lund University, Lund, Sweden